CLINICAL TRIAL: NCT04804345
Title: AProtinin Versus Tranexamic Acid in Cardiac Surgery Patients With High-risk for Excessive Bleeding
Acronym: APACHE
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2020/67
Record Dates: First submitted 2021-03-10; First posted 2021-03-18 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: Cardiac Surgery; Cardiopulmonary Bypass; High Risk Bleeding
Keywords: cardiac surgery; cardiopulmonary bypass; massive peri-operative bleeding; antifibrinolytics; blood products transfusion
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The aprotinin group,: all patients receiving a first infusion 1M KIU before surgical incision followed by a steady dose of 250 000 KIU/h with an additional dose of 1M KIU added to the cardiopulmonary bypass unit.
  Interventions: Other: standard of care
- The tranexamic acid group: all patient receiving tranexamic acid following each local center standarded protocol
  Interventions: Other: standard of care

INTERVENTIONS:
Other: standard of care — retrospective study: standard of care

SUMMARY:
In this before-after multicenter study the authors tested the hypothesis that the prophylactic use of aprotinin compared to tranexamic acid could reduce the proportion of patients presenting severe perioperative bleeding.

DETAILED DESCRIPTION:
Perioperative bleeding remains a real challenge for physicians managing cardiac surgical patients. In patients at high risk for excessive bleeding the prophylactic use of antifibrinolytics may be useful. This study propose to compare the efficacity and innocuity of aprotinin and tranexamic acid to reduce the proportion of patient presenting severe peri-operative bleeding according the Universal Definition of Perioperative Bleeding (UDPB) classification.

ELIGIBILITY:
Inclusion Criteria:

patients undergoing cardiac on pump surgery at high risk for bleeding defined by :

* Aorto-coronary bypasses surgery (2 or more) under dual platelet aggregation therapy (Primary or redo)
* Heart transplant (Primary or Redo)
* Infectious endocarditis (Primary or Redo)
* Ascending acute aortic dissection (Primary or Redo)
* Artificial heart / LVAD under CEC (Primary or Redo)
* Combined surgery, Redo
* Ascending aorta surgery, Redo

Exclusion Criteria:

* Off pump cardiac surgery
* Patient not meeting the inclusion criteria
* Patient not receiving antifibrinolytic therapy
* Patient with absolute contraindication to antifibrinolytics,
* Patient refusing to give access to their medical chart,
* Patient not meeting the inclusion criteria
* Patient protected by the law, under guardianship or trusteeship,
* Patient deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive patients undergoing cardiac surgery with a high risk of hemorrhage who have received a prophylactic infusion of either tranexamic acid or aprotinin and meeting the protocol criteria between july 2017 and october 2020 in seven university hospital centers.
Sampling Method: Probability Sample
Enrollment: 693 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with severe peri-operative bleeding | day 30 after surgery
  Proportion of patients with severe peri-operative bleeding defined by an UDPB (the Universal Definition of Perioperative Bleeding ) classification of 3 and 4.

SECONDARY OUTCOMES:
distribution of patients by UDPB classification category | day 30 after surgery
  proportion of patients with category 0 UDPB.
distribution of patients by UDPB classification category | day 30 after surgery
  proportion of patients with category 1 UDPB.
distribution of patients by UDPB classification category | day 30 after surgery
  proportion of patients with category 2 UDPB.
distribution of patients by UDPB classification category | day 30 after surgery
  proportion of patients with category 3 UDPB.
distribution of patients by UDPB classification category | day 30 after surgery
  proportion of patients with category 4 UDPB.
blood loss | 24 hours after chest closure
  post operative chest tube blood loss
rescue surgery for bleeding | day 30 after surgery
  proportion of rescue surgery for bleeding
length of stay | through intensive care unit discharge, an average of 30 days
  intensive care unit length of stay
length of stay | through hospital discharge, an average of 30 days
  hospital length of stay
KDIGO score greater than or equal to 2 | day 7 after surgery
  acute kidney injury defined by KDIGO score greater than or equal to 2
mechanical ventilation time | through intensive care unit discharge, an average of 30 days
  duration of artificial ventilation (hours)
mechanical ventilation | 48 hours after surgery
  need to use mechanical ventilation for more than 48 hours
need for transfusion | up to 48 hours after surgery
  need for labil blood products and medicinal products derived from blood
need for transfusion | up to seven day after surgery
  need for labil blood products and medicinal products derived from blood
need for vasopressors/inotropes | beyond 24 hours after surgery
  need for use postoperative vasopressors/inotropes for more than 24 hours
vital status | 30 days after surgery
  mortality after surgery
new renal replacement therapy | up to day 30 after surgery
  need for renal replacement therapy
short term mechanical circulatory support | up to 30 day after surgery
  need for short term mechanical circulatory support (extra corporeal life support, Impella TM pump, intra aortic balloon pump)
myocardial infarction | up to 30 day after surgery
  occurrence of myocardial infarction
embolic or thrombotic event | up to 30 day after surgery
  occurrence of embolic or thrombotic event
stroke | up to 30 day after surgery
  occurrence of stroke

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre OUATTARA, MD, PhD, Principal Investigator — University Hospital, Bordeaux
Locations (7):
- France (7):
  - Grenoble University Hospital, La Tronche
  - Lyon University Hospital, Lyon
  - Montpellier University Hospital, Montpellier
  - Nantes University Hospital, Nantes
  - North Val de Seine Paris University Hospital, Paris
  - Georges Pompidou European University Hospital, Paris
  - Bordeaux University Hospital, Pessac

IPD SHARING:
Plan to Share IPD: No